CLINICAL TRIAL: NCT00756912
Title: A Phase I, Open-Label, Dose Escalation Study of Eritoran (E5564) Administered IV Over 14 Days Prior to and During Bone Marrow Engraftment in BMT Patients Who Have Received Myeloablative Conditioning Treatment and Are Receiving Bone Marrow or Stem Cells From Matched Related Donors
Brief Title: A Study of Eritoran (E5564) Administered IV Over 14 Days Prior to and During Bone Marrow Engraftment in BMT Patients Who Have Received Myeloablative Conditioning Treatment and Are Receiving Bone Marrow or Stem Cells From Matched Related Donors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This study was terminated in November 2008 due to "a business decision (resources)".
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: E5564-A001-102
Record Dates: First submitted 2008-09-18; First posted 2008-09-22 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2014-07

CONDITIONS: Leukemia
Keywords: ANC; BMT; graft versus leukemia; graft vs. host disease; MD2 (endotoxin binding-protein); undergo allogeneic BMT; myeloablative; conditioning; therapy
MeSH Terms: conditions — Leukemia; Graft vs Host Disease | interventions — E5564; eritoran

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: E5564

INTERVENTIONS:
Drug: E5564 — Three dose levels of Eritoran IV over 14 days for a total of 32, 96, and 224 mg over 14 days.
  Other Names: Eritoran

SUMMARY:
This is a study designed to assess the safety of administration of up to 3 dose levels of eritoran in subjects undergoing or scheduled to undergo allogeneic bone marrow transplant (BMT). An allogeneic BMT is the transplantation of blood stem cells taken from the bone marrow or blood of another person.

DETAILED DESCRIPTION:
Please note: in the original protocol, the study phase is listed as "Phase Ib", although the Official Title reads "Phase I".

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the inclusion criteria outlined below in order to be eligible to participate in this study:

1. Adult subjects (aged 18 to 55 years old) undergoing or scheduled to undergo myeloablative conditioning and allogeneic BMT, or stem cells from matched donors.
2. Subjects using either busulfan or total body irradiation (TBI) containing regimens for BMT for the treatment of malignant and nonmalignant diseases. For example:

   * Cyclophosphamide and Total Body Irradiation (CY-TBI) with a TBI dose of at least 1200 cGy of fractionated TBI
   * Etoposide and Total Body Irradiation (VP16-TBI) with a TBI dose of at least 1200 cGy of fractionated TBI
   * Busulfan and cyclophosphamide (BU-CY) with at least 14 mg/kg busulfan orally or 11.2 mg/kg busulfan intravenously (14 x 0.8 correction factor) or a targeted busulfan dosing strategy aimed at a serum concentration greater than 600 ng/mL at steady state.
3. Leukemia patients with:

   * acute myelogenous leukemia (AML)
   * acute lymphoblastic leukemia (ALL) in first or subsequent complete remission
   * chronic myelogenous leukemia (CML) in first or subsequent chronic phase or in accelerated phase
   * myelodysplastic syndrome (MDS) patients.

   OR

   Subjects with non-Hodgkin's lymphoma who are in complete remission as determined by physical exam, CT and PET scans, and are otherwise considered candidates for allogeneic BMT as judged by the treating institution
4. Available matched related CD34+ stem cells (target cell dose between 2 x 10^6/kg and 10 x 10^6/kg (actual body weight)) for transplantation (matched at 6/6 HLA at Class I HLA-A and B and Class II HLA-DRBI).
5. Sex distribution: men or nonpregnant women. Women of childbearing potential must have a negative serum β-human chorionic gonadotropin (hCG) or urine assay prior to eritoran treatment or prior to the beginning of conditioning treatment. Menopausal women must have been amenorrheic for at least 12 months.
6. Race: any.
7. Has signed informed consent before any study-specific procedures are performed.

Exclusion Criteria:

1. Unwilling or unable to agree to be fully evaluated for all follow-up visits. The subject or subject's representative and the study staff should agree to perform all study assessments even if the subject is discharged from the hospital.
2. Seropositive for human immunodeficiency virus (HIV); testing is not needed if already performed (documentation required) as part of screening for conditioning treatment.
3. Subjects with a documented or possible systemic infection, or suspected of having a medically significant viral, bacterial, or fungal infection at the beginning of treatment on Day -3.
4. Have taken any investigational medications (ie, not approved by the FDA for any indication) within the 30-day period prior to enrollment into the study.
5. Karnofsky Performance Status (KPS) <60%.
6. Have previously received a bone marrow or stem cell transplant.
7. Are to receive T-cell depleted BMT or stem cell infusions.
8. Are pregnant or lactating.
9. Known sensitivity to eritoran or its excipients.
10. Prior malignancies treated with a curative intent of < 5 years will not be allowed. Previously treated cancer with a curative intent of > 5 years will be allowed.
11. Legal incapacity.
12. Any of the following laboratory parameters within 2 days prior to the beginning of treatment on Day -3:

    * direct bilirubin ≥ 2x ULN
    * liver function tests (ALT or AST) with values ≥ 3x ULN
    * serum creatinine ≥ 2x ULN
13. Subjects who are enrolled in other interventional, investigational protocols. As aGvHD is likely to only occur after treatment with eritoran is completed, investigational treatments for Grades III and IV aGvHD may be allowed and should be discussed with the Sponsor.
14. Subjects with a history of or with current pulmonary disease with forced vital capacity (FVC) or forced expiratory volume in 1 second (FEV1) < 60% predicted (corrected for hemoglobin).
15. Subjects with a history of a cardiac ejection fraction < 45%, or with marked screening or baseline prolongation QT/QTc interval (QTc interval > 470 mSec).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2008-09; Primary Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Safety and assessments will be done daily. | Performed daily through Day 28, with follow-up every other week to Day 100 and at 1 year post-transplant.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Cooke, Principal Investigator — Case Western Reserve University School of Medicine
Locations (1):
- Case Western Reserve University School of Medicine, Cleveland, Ohio, United States